CLINICAL TRIAL: NCT01477541
Title: Incorporation of Alternative Providers for Care During Pregnancy, Delivery and Postpartum in Rural Public Health Clinics.
Brief Title: Cluster-randomized Trial Measuring Integration of Professional Midwives and Obstetric Nurses in Rural Clinics in Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Mexican National Institute for Women (Unknown); Mexican Center for Gender Equity and Reproductive Health (Unknown); Secretary of Health, Guerrero state (Unknown); Secretary of Health, Oaxaca state (Unknown)
Responsible Party: Principal Investigator, Dilys Walker, Investidadora Asociada C, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 104-6466
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Pregnancy
Keywords: Prenatal care; Maternal mortality; Perinatal mortality; Perinatal; Puerperium; Puerperium care; Midwives; Midwife; Obstetric; Nurse; Integration; Alternative personnel; Skilled attendant; Birth attendant; Delivery; Delivery services; Best practices; Rural
MeSH Terms: conditions — Maternal Death; Perinatal Death

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- PM/ON integration arm (Experimental): Health centers where professional midwives or obstetric nurses are integrated into clinic staff and delivering services.
  Interventions: Other: PM/ON integration
- Control (No Intervention)

INTERVENTIONS:
Other: PM/ON integration — Professional midwives or obstetric nurses are integrated into clinic staff and delivering services.
  Arms: PM/ON integration arm

SUMMARY:
Rates and causes of maternal mortality in Mexico have dropped only slightly; thus, reaching the internationally established Millennium Development Milestones (MDM) is still a distant goal. A fundamental part of reducing maternal and infant mortality is ensuring skilled attendance during pregnancy and delivery. This project uses an innovative strategy of integrating professional midwives and licensed obstetric nurses into rural medical centers in the states of Guerrero and Oaxaca, Mexico, to provide prenatal care, delivery services, and puerperium care. The goal of the research is to increase use of best practices in intake, labor, delivery, and puerperium care; decrease the use of unnecessary or harmful care; and improve maternal and neonatal outcomes. We posited that medical centers receiving the intervention would provide better care and have better maternal and neonatal outcomes than those that did not receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinics containing one medical team only (1 doctor and accompanying staff)
* Clinics less than 2 hours away from a referral hospital
* Clinics where at least 25 deliveries took place in the previous year

Exclusion Criteria:

* Clinics inaccessible by car
* Clinics undergoing remodeling

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Use of evidence-based practices during labor, delivery, and postpartum care | 21 months
  Will collect data on deliveries ocurring in sites over 21 month period.
volume of prenatal visits, deliveries | 21 months
  We will Assess overall number of first and follow up prenatal visits and deliveries in intervention and control sites
Use of harmful or unnecessary practices during labor and delivery | 21 months
  We will assess use of harmful or unnecessary practices during labor and delivery

CONTACTS AND LOCATIONS:
Overall Officials: Dilys Walker, MD, Principal Investigator — Instituto Nacional de Salud Publica, Mexico